CLINICAL TRIAL: NCT01124396
Title: A Double-blind, Placebo-controlled, Randomised Study to Investigate the Tolerability, Safety, Pharmacokinetics and Pharmacodynamics of Repeated Weekly Doses of DSP-3025 Administered Intranasally to Healthy Male Volunteers
Brief Title: DSP-3025 A Phase 1 Study of Healthy Male Volunteers
Status: Completed | Type: Observational
Sponsor: Sumitomo Pharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: D7002027
Record Dates: First submitted 2010-05-13; First posted 2010-05-17 (Estimated); Last update posted 2022-04-12 (Actual); Status verified 2022-04

CONDITIONS: Healthy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (3):
- 30 ug: 30 ug
  Interventions: Drug: DSP-3025
- 60 ug: 60 ug
  Interventions: Drug: Placebo
- Placebo: Placebo

INTERVENTIONS:
Drug: DSP-3025
  Groups: 30 ug
Drug: Placebo
  Groups: 60 ug

SUMMARY:
Investigate safety/tolerability after repeated weekly doses intranasal administration of DSP-3025 comparator placebo to healthy male volunteers

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) between 18.5 and 25 kg/ m2 and a weight between 50 and 80 kg
* No clinically relevant abnormal findings

Exclusion Criteria:

* Acute illness which requires medical intervention
* Definite or suspected personal history of adverse drug reactions or drug hypersensitivity
* Clinical relevant disease or disorder (past or present)
* A history of respiratory disorder(s) such as asthma

Ages: 20 Years to 39 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Sampling Method: Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2010-04; Primary Completion 2010-08 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Incidence/nature of adverse events, 12-lead ECG, pulse, BP, body temperature, spirometry | During the study

SECONDARY OUTCOMES:
Clinical chemistry, haematology, urinalysis, autoantibodies | During the study
Nasal symptoms and peak nasal inspiratory flow | During the study
Pharmacokinetics | During the study
Biomarkers nasal lavage and blood | During the study

CONTACTS AND LOCATIONS:
Locations (1):
- Kitasato University East Hospital, Asamizodai 2-1-1, Minami-ku, Sagamihara, Kanagawa, Japan